CLINICAL TRIAL: NCT06303011
Title: Effects of Abdominal Massage With TENS on Para Sacral Versus Sacral Area on Symptom Severity and Quality of Life in Severe Chronic Constipation Among Young Females
Brief Title: Abdominal Massage With TENS on Parasacral Versus Sacral Area on Symptom,Severity & QOL in Chronic Constipation Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S22C14G92003
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Constipation
Keywords: Constipation; Quality of life; Abdominal massage
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group: A (Experimental): TENS on sacral areas with Abdominal Massage
  Interventions: Other: Transcutaneous Electrical Nerve Stimulator
- Group: B (Active Comparator): TENS on para sacral area with Abdominal Massage
  Interventions: Other: TENS on para sacral area with Abdominal Massage

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulator — TENS will be applied on sacral and parasacral area. Frequency 10Hz, Pulse duration 200μs, Stimulation duration 20min
  Arms: Group: A
Other: TENS on para sacral area with Abdominal Massage — TENS on para sacral area with Abdominal Massage. Frequency 10Hz Pulse duration 200μs Stimulation duration 20min
  Arms: Group: B

SUMMARY:
Constipation is Infrequent or difficult evacuation of FECES. These symptoms are associated with a variety of causes, including low DIETARY FIBER intake, emotional or nervous disturbances, systemic and structural disorders, drug-induced aggravation, and infections. Patients complaining of constipation may mean different things by the term The frequency of their bowel actions may be less than 'normal', their stools maybe difficult to pass, or they may have a sense of malaise or abdominal discomfort which they attribute to a 'sluggish bowel', though the stool frequency and consistency are apparently normal. Objective of this study is to compare effects of Abdominal massage. withTENSonparasacralversussacralareaonsymptomseverityandqualityoflifein severechronicconstipationamongyoungfemales.

DETAILED DESCRIPTION:
This study will be a Randomized Clinical trial and will be conducted at services Hospital in Lahore. The study will be completed with in the time duration of eight months. Purposive sampling technique will be used to collect the data. A sample size of Total 24 patients will be taken in this study. Patients will be divided into two groups.(Group A will be treated with TENS on sacral area and abdominal massage where as Group B will be treated with TENS on par sacral area and abdominal massage).PAC-SYM Questionaire,PAC-QOL Questionaire will be used to ask some questions related to patients 'symptoms and abdominal cramps or bloating.. All participants of the study will fill the PAC-SYMQ and PAC-QOL Q on day 1 as pre treatment values and at the end of 4th session as post treatment values respectively. The collected data will be analyzed on SPSS-25.

Keywords : constipation, Quality of life , abdominal massage.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 -35year
* Only females
* Laxatives at least once or more for 2weeks
* Non pregnant
* Chronic Constipation more then 6 months

Exclusion Criteria:

* Organic dysphasia or secondary constipation caused by laxatives for unrelated conditions.
* Pregnant females suspected pregnant subjects, as well as those who were breast-feeding
* Non co-operative patients
* Female with underlying disease

Ages: 14 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Females experience more constipation
Enrollment: 26 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
PAC-SYM Questionnaire | 8 weeks
  It is a self-reported questionnaire consisting of 12 symptoms divided into three domains: abdominal, rectal and stool, with responses rated on a. 5-point.The Patient Assessment of Constipation-Symptoms (PAC-SYM) questionnaire is frequently used in clinical trials of constipation. However, the threshold for reduction in total PAC-SYM score used to define a clinical response on this 0-4 point scale has not undergone formal appraisal, and its relationship with clinical benefit as perceived by patients has not been defined.
  PAC-SYM Questionnaire Validity is 0.68 to 0.72 and reliability is 0.75to 0.89
PAC-QOL Questionnaire | 8 weeks
  The following questions are designed to measure the impact constipation has had on your daily life over the past 2 weeks. The overall PAC-QOL score consisted of four domains: physical discomfort, psycho- social discomfort, satisfaction, and worries and concerns. A lower score indicated a better outcome for symptomatic relief and QOL. PAC-QOL Questionnaire Validity is 0.76 to 3.41 and reliability is >0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Taufiq, PPDPT, Principal Investigator — Riphah International University, Senior Lecturer
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No